CLINICAL TRIAL: NCT02814305
Title: Opioid Analgesic Use and Disposal Following Outpatient Dental Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 821823
Record Dates: First submitted 2016-06-16; First posted 2016-06-27 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Opioid Use Disorders; Tooth Extraction Status Nos
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (4):
- Control (No Intervention): Patient receives neither educational nor financial interventions
- Financial intervention only (Experimental): Patient receives financial (pharmacy offer) intervention only
  Interventions: Behavioral: Financial
- Educational intervention only (Experimental): Patient receives educational (narrative) intervention only
  Interventions: Behavioral: Educational
- Both interventions (Experimental): Patient receives both educational and financial interventions
  Interventions: Behavioral: Financial; Behavioral: Educational

INTERVENTIONS:
Behavioral: Financial — Patient receives information on a program that may offer a financial benefit for disposing of unused opioid analgesics at a pharmacy
  Arms: Both interventions; Financial intervention only
Behavioral: Educational — Patient watches a video featuring narrative vignettes of patients who developed opioid dependence or abuse after using opioids postoperatively
  Arms: Both interventions; Educational intervention only

SUMMARY:
Background: Overdose deaths from prescription opioid analgesics quadrupled from 4,000 cases to nearly 17,000 cases annually during 1999-2011. Most people who misuse or abuse prescription opioids obtain these pills from friends or family members who have surplus medication left over from prior prescriptions. There is little published data on surplus opioid analgesics remaining after patients recover from painful procedures. Even less is known about patients' willingness to dispose of these leftover pills.

Aims: 1) Measure the impact of a risk education intervention and a financial incentive intervention on patients' willingness to dispose of surplus opioids left over after outpatient dental surgery. 2) Measure the number and proportion of opioid pills left unused after outpatient dental surgery.

Methods: The study will be a pilot randomized controlled trial. Adult patients at the Penn Dental Care Center will be enrolled prior to elective outpatient dental surgery. Patients will be randomized to a control group, an educational intervention, or a financial incentive intervention. The primary outcome of the trial is the proportion of patients in each arm that express willingness to return their unused opioids. Secondary outcomes include patient use of prescribed opioids and their number of unused pills. These outcomes will be measured using novel text-message based data collection software that patients will interact with using a web-enabled cellular telephone or tablet.

ELIGIBILITY:
Inclusion Criteria:

* Non-institutionalized

Exclusion Criteria:

* pregnancy
* a history of opioid analgesic misuse/abuse
* ongoing participation in other clinical research
* or daily use of opioid analgesics in the week prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2015-03; Primary Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Unused opioids | 21 days after surgery
  Number of opioids reported unused by the patient after postoperative day 21

SECONDARY OUTCOMES:
Intent to dispose of opioids | Any time during the 21-day data collection period or during the follow-up interview on (or shortly after) postoperative day 21
  Patient reports intent to dispose of leftover opioids during follow-up interview or by calling study hotline